CLINICAL TRIAL: NCT04515082
Title: Colorectal Cancer and Advanced Precancerous Neoplasm Screening Using Stool DNA-based SDC2 and SFRP2 Methylation Test in China, a Multi-Center Study
Brief Title: Colorectal Cancer Screening Using Stool DNA-based SDC2 and SFRP2 Methylation Test in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, MD, Director, Head of Department of Gastroenterology and Digestive Endoscopy Center, Principal Investigator, Clinical Professor, Changhai Hospital
Other Study IDs: CHEC2020-033
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Neoplasm; Colorectal Cancer; Adenomatous Polyps; Adenoma; Advanced Adenoma; Serrated Polyp
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyps; Adenoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stool-based SDC2 and SFRP2 DNA methylation test — A diagnostic device measuring syndecan 2 (SDC2) and secreted frizzled-related protein 2 (SFRP2) methylation status in stool DNA to detect colorectal cancer
  Other Names: Colowell
Diagnostic Test: FIT — Fecal immunochemical test

SUMMARY:
The primary objective is to determine sensitivity, specificity, positive predictive value and negative predictive value of a bi-target stool DNA testing (the methylation status of SDC2 and SFRP2) for colorectal cancer and advanced precancerous neoplasm(including advanced adenoma and advanced serrated lesions) screening, using colonoscopy as the reference method. Lesions will be confirmed as malignant or precancerous by histopathologic examination.

The secondary objective is to compare the performance of the bi-target stool DNA testing to a commercially available fecal immunochemical test (FIT) assay, both with respect to cancer and advanced precancerous neoplasm. Lesions will be confirmed as malignant or precancerous by colonoscopy and histopathologic examination.

DETAILED DESCRIPTION:
This study is a multi-center diagnostic test led by the National Clinical Research Center for Digestive Disease (Shanghai) (Department of Gastroenterology, Changhai Hospital, Navy/Second Military Medical University), which is conducted at about 30 digestive endoscopy centers nationwide in China, with the expectation of including approximately 4,800 patients. Subjects willing to conduct colonoscopy examination will be asked to collect stool sample prior to bowl preparation for stool DNA test and commercially available FIT assay. The basic characteristics of subjects, bowel preparation method and quality, and related information of colonoscopy are recorded in detail. Colonoscopy and histopathologic examination are used as reference.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 to 85 years old, the gender is not limited
2. Willing to provide written consent
3. Able to provide stool sample

Exclusion Criteria:

1. Unwilling to provide stool samples
2. Subject with contraindications for bowel preparation or colonoscopy
3. Subject with known colorectal polyps but not removed
4. Subject with inflammatory bowel disease
5. History of colonoscopy within 1 year
6. History of colorectal cancer
7. History of hereditary colorectal cancer syndrome (including polyposis)
8. Active lower gastrointestinal bleeding
9. Pregnancy
10. Subject taking anticoagulants such as aspirin and warfarin, or who have coagulopathy
11. Subject clinically highly suspected with gastrointestinal cancer
12. Other conditions deemed not suited for the study by investigators

Elimination Criteria:

1. Ask to withdraw from the study
2. Unable to get a stool sample
3. Invalid stool samples to test
4. Poor or inadequate bowel preparation
5. Failed to complete the colonoscopy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who referred to the outpatient and received colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value of bi-target stool DNA testing (the methylation status of SDC2 and SFRP2) with comparison to colonoscopy, both with respect to cancer and advanced precancerous neoplasm. | Through study completion, an average of 1 year
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant or precancerous by histopathologic examination. Advanced precancerous neoplasm includes both advanced adenoma and advanced serrated lesions. The DNA test includes the methylation status of SDC2 and SFRP2. The tests were processed independently of colonoscopy procedure.

SECONDARY OUTCOMES:
To compare the performance of the bi-target stool DNA testing to a commercially available FIT assay, both with respect to cancer and advanced precancerous neoplasm. | Through study completion, an average of 1 year
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant or precancerous by histopathologic examination. The stool DNA and FIT test were performed on the same stool sample.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital, Navy/Second Military Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niu F, Wen J, Fu X, Li C, Zhao R, Wu S, Yu H, Liu X, Zhao X, Liu S, Wang X, Wang J, Zou H. Stool DNA Test of Methylated Syndecan-2 for the Early Detection of Colorectal Neoplasia. Cancer Epidemiol Biomarkers Prev. 2017 Sep;26(9):1411-1419. doi: 10.1158/1055-9965.EPI-17-0153. Epub 2017 Jun 15. PMID 28619831
- [Background] Oh TJ, Oh HI, Seo YY, Jeong D, Kim C, Kang HW, Han YD, Chung HC, Kim NK, An S. Feasibility of quantifying SDC2 methylation in stool DNA for early detection of colorectal cancer. Clin Epigenetics. 2017 Dec 4;9:126. doi: 10.1186/s13148-017-0426-3. eCollection 2017. PMID 29225717
- [Background] Han YD, Oh TJ, Chung TH, Jang HW, Kim YN, An S, Kim NK. Early detection of colorectal cancer based on presence of methylated syndecan-2 (SDC2) in stool DNA. Clin Epigenetics. 2019 Mar 15;11(1):51. doi: 10.1186/s13148-019-0642-0. PMID 30876480
- [Background] Huang Z, Li L, Wang J. Hypermethylation of SFRP2 as a potential marker for stool-based detection of colorectal cancer and precancerous lesions. Dig Dis Sci. 2007 Sep;52(9):2287-91. doi: 10.1007/s10620-007-9755-y. Epub 2007 Apr 5. PMID 17410438
- [Background] Oberwalder M, Zitt M, Wontner C, Fiegl H, Goebel G, Zitt M, Kohle O, Muhlmann G, Ofner D, Margreiter R, Muller HM. SFRP2 methylation in fecal DNA--a marker for colorectal polyps. Int J Colorectal Dis. 2008 Jan;23(1):15-9. doi: 10.1007/s00384-007-0355-2. Epub 2007 Jul 17. PMID 17639423
- [Background] Wang DR, Tang D. Hypermethylated SFRP2 gene in fecal DNA is a high potential biomarker for colorectal cancer noninvasive screening. World J Gastroenterol. 2008 Jan 28;14(4):524-31. doi: 10.3748/wjg.14.524. PMID 18203283
- [Background] Zhou Z, Zhang H, Lei Y. Diagnostic value of secreted frizzled-related protein 2 gene promoter hypermethylation in stool for colorectal cancer: A meta-analysis. J Cancer Res Ther. 2016 Oct;12(Supplement):30-33. doi: 10.4103/0973-1482.191625. PMID 27721248